CLINICAL TRIAL: NCT07177131
Title: Prospective, Randomized Cross-over Within-subject Study on the Effects of Dehydration and Hyperhydration on Macular Thickness, Corneal Morphology, and Ocular Biometric Parameters Measured by OCT, Pentacam and Optical Biometer
Brief Title: Hydration Status and Ocular Parameters Study
Acronym: HYDRI-EYE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ante Kreso (Other)
Collaborators: University Hospital of Split (Other); University of Split, School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Ante Kreso, Principal Investigator, University Hospital of Split
Organization: University Hospital of Split (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: JC092025
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hydration Status; Macular Thickness; Ocular Biometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relative Dehydration (Experimental): 12-hour fluid restriction (≤250 ml fluids until 20h previous day)
  Interventions: Behavioral: Relative Dehydration Protocol
- Hyperhydration (Experimental): 2 liters of water within 4 hours before testing
  Interventions: Behavioral: Hyperhydration Protocol

INTERVENTIONS:
Behavioral: Relative Dehydration Protocol — Participants will abstain from water intake for 12 hours prior to the study visit. Food is allowed, but fluid intake is limited to a maximum of 250 ml until 20:00 h on the previous evening. Eye measurements will be performed in the morning (8-10 h).
  Arms: Relative Dehydration
Behavioral: Hyperhydration Protocol — Participants will consume 2 liters of water within 4 hours prior to the study visit. Eye measurements will be performed in the morning (8-10 h).
  Arms: Hyperhydration

SUMMARY:
This study will examine how hydration status (drinking a large amount of water or avoiding water for a short period of time) affects the eye. Healthy adult volunteers will participate in two sessions: one after mild dehydration (no water for 12 hours) and one after drinking 2 liters of water within 4 hours. At each session, detailed eye measurements will be taken, including scans of the retina and optic nerve using optical coherence tomography (OCT), corneal imaging with Pentacam, and eye length measurements with an optical biometer. The results from the two conditions will be compared within the same participants.

The main goal is to determine whether hydration influences the thickness of the retina (macula). Secondary goals include assessing changes in the optic nerve, cornea, and other biometric eye parameters. The study involves only non-invasive tests and minimal risk. Findings may help improve understanding of how hydration affects the eye and may be important for clinical practice, such as planning cataract or refractive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 18 to 65 years
* Normal ophthalmological findings
* Best corrected visual acuity (BCVA) ≥ 1.0 (decimal)
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Known ocular diseases (e.g., glaucoma, keratoconus, retinal pathology)
* History of ocular surgery
* Systemic diseases affecting hydration status (e.g., diabetes mellitus, kidney disease)
* Any condition that, in the investigator's opinion, could interfere with study participation or data quality
* Refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in macular thickness between dehydration and hyperhydration states | Within 1 week (cross-over design with ≥7-day washout period)
  Macular thickness (central subfield, parafoveal, and perifoveal regions) will be measured using Zeiss Cirrus HD-OCT. Each participant will undergo measurements in both hydration states, and paired comparisons will be performed.

IPD SHARING:
Plan to Share IPD: Undecided